CLINICAL TRIAL: NCT02537041
Title: Non-invasive Evaluation of Myocardial Stiffness by Elastography in the Elderly Suffering From Isolated Diastolic Heart Failure: New Diagnostic Tool?
Brief Title: Non-invasive Evaluation of Myocardial Stiffness by Elastography
Acronym: Elasto-Cardio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: French Cardiology Society (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-02
Record Dates: First submitted 2015-08-24; First posted 2015-09-01 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Diastolic Heart Failure
MeSH Terms: conditions — Heart Failure, Diastolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- healthy volunteers (Other): to obtain normal values diastolic myocardial stiffness references. The objective will be to confirm the increase with age in myocardial stiffness assessed by elastography in healthy subjects.
  Interventions: Procedure: elastography function ShearWave Imaging; Procedure: MRI
- diastolic Heart Failure (Other): older patients with isolated diastolic HF (EF> 45%, 60-80 years, n = 20) and infiltrative cardiomyopathy restrictive-type amyloidosis (n = 20) . The objective will be to study the results of elastography on two separate clinical types of IC diastolic well identified.
  Interventions: Procedure: elastography function ShearWave Imaging; Procedure: MRI
- systolic Heart Failure (Other): elderly patients with heart failure with impaired ejection (<45%) fraction, but no segmental dysfunction.
  The evaluation of myocardial stiffness by elastography in all these patients will be compared to conventionally ultrasound and biological parameters currently used for diagnosis of elderly's diastolic HF
  Interventions: Procedure: elastography function ShearWave Imaging; Procedure: MRI

INTERVENTIONS:
Procedure: elastography function ShearWave Imaging — non-invasive assessment of myocardial stiffness by elastography
Procedure: MRI

SUMMARY:
SITUATION ON RESEARCH Diastolic heart failure (HF) or heart failure with preserved systolic function (SF) is the primary cause of heart failure in the elderly (over 2/3 of heart failure in patients over 60 years). Its main cause is hypertension. The diagnosis of diastolic heart failure is still controversial in clinical practice. It is based on ultrasound and biological criteria (or MRI). Basically, it is concerned patients making acute pulmonary edema with preserved SF and high BNP. It is now recognized that the "primum movens" of this type of HF is increased myocardial stiffness secondary to LVH. Noninvasive assessment of this parameter would allow a more accurate and reliable diagnosis because not dependent on load conditions unlike the ejection fraction (EF) and trans-mitral Doppler. However, the absence of non-invasive tool for the direct evaluation of the diastolic stiffness (so-called passive) prevents to date to use this diagnostic parameter.

The investigators propose here to evaluate noninvasively myocardial stiffness in elderly patients with diastolic heart failure using a new imaging tool that uses an innovative ultrasonic technology, the ultrafast echo associated with its elastography function "ShearWave Imaging" (SWI). The investigators work for several years in collaboration with the Langevin Institute on this technology which was recently validated in experimental models. Its principle is based on the creation of a shear wave from a standard ultrasound and calculating the velocity of this wave with the high time resolution of the ultrasound probe, this being correlated with the speed myocardial stiffness.

The human study was recently made possible by the development of a phased array probe having the opportunity to work with elastography mode (SWI).

PURPOSE OF RESEARCH The goal will be to demonstrate the interest of the non-invasive evaluation by ultrafast echo (SWI) of myocardial stiffness in the diagnosis of diastolic heart failure in the elderly.

DETAILED DESCRIPTION:
DESCRIPTION PROJECT SUMMARY

Three groups of patients in sinus rhythm will be studied (n total = 100 patients):

* Group 1 "healthy volunteers" (n = 40): two age classes determined ([20-40ans, n = 20] and [60-80 years, n = 20]), to obtain normal values diastolic myocardial stiffness references. The objective will be to confirm the increase with age in myocardial stiffness assessed by elastography in healthy subjects.
* Group 2 "diastolic HF" (n = 40): older patients with isolated diastolic HF (EF> 45%, 60-80 years, n = 20) and infiltrative cardiomyopathy restrictive-type amyloidosis (n = 20) . The objective will be to study the results of elastography on two separate clinical types of IC diastolic well identified.
* Group 3 "systolic HF" (n = 20): elderly patients with heart failure with impaired ejection (<45%) fraction, but no segmental dysfunction.

The evaluation of myocardial stiffness by elastography in all these patients will be compared to conventionally ultrasound and biological parameters currently used for diagnosis of elderly's diastolic HF. Our hypothesis is that myocardial stiffness assessed by SWI is a powerful parameter for predicting diastolic heart failure. To this end, a univariate and multivariate statistical analysis will be carried out from all of these data.

EXPECTED RESULTS AND OUTLOOK The current ultrasound diagnostic parameters of diastolic heart failure (ESC 2012) using Doppler (trans-mitral tissue) anatomical, or functional (strain, strain rate, speckle tracking) criteria that are dependent on load conditions and are not specific to diastolic HF. This study should demonstrate the continuity of our preclinical studies, the non-invasive assessment of myocardial stiffness by elastography is a powerful test for the detection and diagnosis of diastolic heart failure. Secondly the prognosis character of recovery rates will be studied over a large population of people with HF and FE preserved (diastolic HF) with longitudinal follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 "healthy volunteers" (n = 40): two age classes determined ([20-40ans, n = 20] and [60-80 years, n = 20]),
* Group 2 "diastolic HF" (n = 40): older patients with isolated diastolic HF (EF> 45%, 60-80 years, n = 20) and infiltrative cardiomyopathy restrictive-type amyloidosis (n = 20)
* Group 3 "systolic HF" (n = 20): elderly patients with heart failure with impaired ejection (<45%) fraction, but no segmental dysfunction

Exclusion Criteria:

* pregnant woman
* atrial fibrillation
* patient with defibrillator, pacemaker
* contraindication to MRI
* no consent form
* echography gel allergy
* participation to another study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-09; Primary Completion 2017-03 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
myocardial stiffness ( measured by kPa) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Olivier VILLEMAIN, MD, Study Chair — LAngevin Institute
Locations (1):
- Hopital Europeen Georges Pompidou, Paris, France

REFERENCES:
- [Derived] Villemain O, Correia M, Mousseaux E, Baranger J, Zarka S, Podetti I, Soulat G, Damy T, Hagege A, Tanter M, Pernot M, Messas E. Myocardial Stiffness Evaluation Using Noninvasive Shear Wave Imaging in Healthy and Hypertrophic Cardiomyopathic Adults. JACC Cardiovasc Imaging. 2019 Jul;12(7 Pt 1):1135-1145. doi: 10.1016/j.jcmg.2018.02.002. Epub 2018 Mar 14. PMID 29550319